CLINICAL TRIAL: NCT04608812
Title: A Pilot Study of Intratumorally and Intraparenchymally Administered OS2966 Using Convection-enhanced Delivery in Patients With Recurrent/Progressive High-grade Glioma Undergoing a Clinically-indicated Surgical Resection
Brief Title: Convection-enhanced Delivery of OS2966 for Patients With High-grade Glioma Undergoing a Surgical Resection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment and financial constraints.
Sponsor: OncoSynergy, Inc. (Industry)
Collaborators: Infuseon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS2966CED-001
Record Dates: First submitted 2020-10-21; First posted 2020-10-29 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Glioma, Malignant; High Grade Glioma; Glioblastoma; Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: CED; Convection-enhanced delivery; recurrent glioblastoma; recurrent high grade glioma; immunotherapy
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma | interventions — gadoteridol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Direct Infusion of OS2966 (Experimental): OS2966 will be directly infused into the brain tumor and surrounding tumor infiltrated brain via convection-enhanced delivery
  Interventions: Drug: OS2966; Drug: Gadoteridol

INTERVENTIONS:
Drug: OS2966 — OS2966 is a humanized monoclonal antibody antagonizing CD29 (Beta 1 integrin)
Drug: Gadoteridol — Gadoteridol is a contrast agent which will be added to OS2966 to allow investigators to observe how OS2966 distributes within the brain tumor. Gadoteridol is approved by the FDA for intravenous injection during an MRI scan. It is not approved by the FDA for administration directly into a tumor.

SUMMARY:
The primary goal of this Phase 1 study is to determine if a new investigational drug, OS2966, when delivered directly to the brain of adult participants with recurrent/progressive high-grade glioma (HGG) is safe and well tolerated.

OS2966 is a therapeutic antibody blocking a cell surface receptor governing fundamental biological processes that allow cancer cells to grow, spread and become resistant to cancer treatment. Despite availability of new promising cancer treatments, successful treatment of HGG has been limited by the presence of the brain's protective blood brain barrier (BBB). The BBB is made up of tightly knit cells that block entry of several substances including cancer treatments. To overcome this obstacle, a technique called convection-enhanced-delivery (CED) will be utilized to deliver OS2966 directly to the site of disease. Convection-enhanced delivery involves placement of one or more catheters into the brain tumor and tumor-infiltrated brain in order to slowly pump a therapy into the tissue.

To be eligible for this study participants must require surgical resection of their recurrent HGG.

DETAILED DESCRIPTION:
This study is an open-label, ascending-dose, 2-part study designed to determine the safety and tolerability of OS2966, as well as the optimal infusion parameters when administering OS2966 directly to the tumor and the surrounding tumor-infiltrated brain by CED in participants with recurrent/progressive HGG undergoing a surgical resection.

OS2966 is an anti-CD29 (Beta1 Integrin) monoclonal antibody (mAb) that has demonstrated preclinical efficacy in resistant/recurrent glioblastoma animal models. This study will recruit participants with recurrent/progressive high-grade glioma (HGG; WHO Grade III or IV glioma). The development of effective treatments for HGG has been limited by an infiltrative growth pattern, the blood brain barrier (BBB), and the rapid development of therapeutic resistance.

Convection-enhanced delivery is a specific technique that allows direct delivery of therapeutics to the brain and to brain tumors. Convection-enhanced delivery bypasses the BBB and allows for infusion of therapeutics that would otherwise be excluded from the central nervous system. Importantly, CEDs targeted delivery obviates systemic toxicity.

Participants enrolled in this study will undergo 2 staged parts of treatment. In Study Part 1, participants will receive a single intratumoral infusion of OS2966 directly to the contrast-enhancing bulk tumor by CED over 4 hours or until maximal tumor coverage is obtained. In Study Part 2, participants will undergo surgical resection of the previously infused tumor. Immediately following surgical resection, catheters will be placed directly into the surrounding tumor-infiltrated brain, and OS2966 will be infused over a 4 hour period and then the catheters removed. To confirm the quality of OS2966 delivery, a gadolinium contrast agent will be added to OS2966 before each infusion in order to monitor the infusion via magnetic resonance imaging.

All participants will be closely monitored clinically, and through the use of imaging assessments to determine how effective OS2966 is at preventing further disease progression. Tumor tissue will be collected in both study parts to evaluate how well OS2966 binds to its intended target and to confirm mechanism of action. All enrolled patients will also receive standard supportive care therapy.

ELIGIBILITY:
Inclusion Criteria

1. Male and female patients aged ≥ 18 years with histologically confirmed diagnosis of a stereotactically accessible, supratentorial, contrast-enhancing WHO Grade III or IV glioma (HGG) with a maximum volume between 2 and 20 cm3.

   • NOTE: Only patients with a histologically confirmed diagnosis of WHO Grade IV glioma (glioblastoma) meeting the above criteria will be eligible for enrollment in the first 3 dose cohorts (ie, dose concentration levels).
2. Patient must have completed standard of care chemoradiation (ie, treatment with temozolomide and radiation) and have evidence of tumor recurrence or progression based on imaging studies within the previous 21 days that supports a clinically-indicated resection.
3. Patient understands the procedures and investigational nature of the study drug and agrees to comply with study requirements by providing written informed consent.
4. Patient must have KPS ≥ 70.
5. At the time of study treatment, patients must have recovered from the toxic effects of prior therapy or meet the following criteria, or both:

   * More than 1 week from last noncytotoxic therapy
   * More than 4 weeks from last cytotoxic therapy, radiation, or treatment with bevacizumab
6. Patient must have adequate bone marrow and organ function as follows:

   a. Adequate bone marrow function:
   * Absolute neutrophil count (ANC) ≥ 1500 μL
   * Leukocyte count ≥ 3000 μL
   * Hemoglobin ≥ 10 g/dL
   * Platelet count ≥ 100,000 μL b. Adequate hepatic function:
   * Aspartate aminotransferase (AST) < 2.5 × institutional upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) < 2.5 × institutional ULN
   * Total bilirubin ≤ 1.5 institutional ULN c. Adequate renal function:
   * Glomerular filtration rate (GFR) ≥ 50 mL/min by Cockcroft Gault equation d. Adequate coagulation function:
   * Prothrombin time (PT)/partial thromboplastin time (PTT) not above institutional norms. Note: patients receiving anticoagulant therapy are eligible for enrollment but must have values below the ULN at the time of surgery.
7. Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control) before study entry, for the duration of the study, and for a minimum of 6 months after study completion.
8. Women of child-bearing potential must have a negative beta-human chorionic gonadoptropin (hCG) serum pregnancy test within 21 days, and a negative urine pregnancy test within 24 hours, before receiving study treatment.
9. Patients must be able to undergo contrast and noncontrast MRI studies.

   Exclusion Criteria

   A patient who meets any of the following criteria will be excluded from participation in this study:
10. Patient has any significant medical illness that, in the investigator's opinion, may compromise the patient's ability to participate in the study.
11. Patient has participated in another investigational therapeutic drug study in the previous 4 weeks.
12. Patient has any of the following tumor characteristics:

    * Multicentric disease - defined as tumors that have multiple discrete areas of contrast enhancement separated by intervening brain and not connected by T2-weighted-Fluid- attenuated Inversion Recovery (FLAIR) abnormality
    * Contrast-enhancing tumor that extends into the opposite cerebral hemisphere
    * Nonparenchymal tumor dissemination (subependymal or leptomeningeal)
    * Tumor located in the posterior fossa
    * Significant mass effect requiring urgent resection.
13. Patient has a history of hypersensitivity reaction to gadolinium contrast agents.
14. Patient is unable to undergo MRI.
15. Patient has a known history of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS).
16. Patient has an active infection (requiring treatment) or an unexplained febrile illness.
17. Patient is receiving anticoagulants, antiplatelets, or nonsteroidal anti-inflammatory drugs (NSAIDs) that cannot be stopped for surgery.
18. Patient is receiving escalating doses of steroids to treat mass effect. Note: patients on stable corticosteroid doses ≤ 4 mg of dexamethasone (or the equivalent of another corticosteroid) daily are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Number of qualifying treatment emergent adverse events or dose limiting toxicities | 28 days
Optimal Biological Dose | 12 months
  Estimated as described in the dosing protocols (accelerated titration and standard 3+3 dose-escalation design).

SECONDARY OUTCOMES:
Spatial Distribution of OS2966 when delivered via CED | Up to 48 hours pre-infusion and up to 24 hours post-infusion
  measured by comparing pre-infusion MR imaging to post-infusion MR Imaging
Tumor Response Rate | 12 months
  based upon MR imaging using RANO criteria assessed every 8 weeks after the initial safety follow up.
Time to Progression | Until progression of disease up to 12 months from infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States